CLINICAL TRIAL: NCT01811251
Title: Co-analgesic Effects of Dexamethasone and Pregabalin After Lumbar Slipped Disc Surgery
Acronym: DEXA-PG-HD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0132; 2012-003157-29
Record Dates: First submitted 2012-12-04; First posted 2013-03-14 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2017-11

CONDITIONS: Patients Undergoing a Lumbar Slipped Disc Surgery
Keywords: Co-analgesia; Dexamethasone; Pregabalin; Lumbar slipped disc surgery; Post-operative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Pregabaline (150mg), Dexamethasone (20mg/5ml; 0.2mg/kg) (Experimental): The aim of the study is to show a decrease in postoperative pain during the first postoperative mobilization surgery lumbar disc herniation through a co-analgesia with a single dose of dexamethasone, pregabalin, or a combination of these two products
  Interventions: Drug: Pregabaline (150mg), Dexamethasone (20mg/5ml; 0.2mg/kg)
- Lactose (150mg), NaC1 0.9% (50ml) (Placebo Comparator): The aim of the study is to show a decrease in postoperative pain during the first postoperative mobilization surgery lumbar disc herniation through a co-analgesia with a single dose of dexamethasone, pregabalin, or a combination of these two products
  Interventions: Drug: Pregabaline (150mg), Dexamethasone (20mg/5ml; 0.2mg/kg)

INTERVENTIONS:
Drug: Pregabaline (150mg), Dexamethasone (20mg/5ml; 0.2mg/kg)

SUMMARY:
The aim of the study is to show a decrease in postoperative pain during the first postoperative mobilization surgery lumbar disc herniation through a co-analgesia with a single dose of dexamethasone, pregabalin, or a combination of these two products.

Pain assessed by simple numerical scale will be also evaluated during the 48 first post-operative hours.

Determining an optimal co-analgesic protocol through the results of this study could help develop validation studies with larger scale such as a medico-economic component. In addition, these study protocols are easy to apply (ponctual administration) and inexpensive.

DETAILED DESCRIPTION:
Visit 1 (J-30 J-1): pre-inclusion visit During a follow-up visit usual pathology, the doctor will propose to the patient to participate in the protocol. Information Form will be given to the patient to be read at home to maintain a sufficient time for reflection. Physician investigator check the eligibility criteria and complete a pre-screening form where he will note the following information about the patient: No pre-enrollment, name, date, reason for non-inclusion appropriate.

Visit 2 (J-1): pre-anesthetic visit, the day before surgery During the pre-anesthetic routine consultation, the doctor will check the proper collection of informed consent and then inform the following information on the CRF: randomization number, age, height, weight, ideal weight theory, gender patient.

Visit 3 (J0): surgery One hour before surgery, the patient will receive, according to randomization, premedication with pregabalin LYRICA ® or placebo orally.

Then the patient will be conducted in the operating room for induction of general anesthesia and surgery. Immediately after induction of anesthesia, depending on randomization, the patient will receive intravenous dexamethasone or placebo.

At the end of surgery, the patient is conducted in Post Anaesthesia Carry Unit (PACU) to be extubated and receive routine care after surgery.

Extubation of the patient, denoted H0 represents the time when the measurement begins.

The data collected from H0 are :

* ENS score standing at H0, H0+30mn, H0+1h, H0+1h30, H0+2 h, H0+6 h,H0+12 h, H0+24h, H0+48 h.
* ENS score mobilization at the first time the patient gets up (edge of the bed and standing if possible)
* Qualification of the quality of standing 0-4 (Likert scale (0 = very poor, 1 = poor, 2 = fair, 3 = good, 4 = very good)) by the nursing staff after the first mobilization
* Qualification of patient satisfaction compared to the first standing by a score of 0-4 (Likert scale (0 = very poor, 1 = poor, 2 = fair, 3 = good, 4 = very good))
* Sedation score at the end of SSPI, , at H0+24h and H0+48h
* Nausea and vomiting score at H0+24 h, H0+48 h
* Tolerance of the treatments undertaken : visual disturbances, lightheadedness, urinary retention, pruritus, measured at the end of SSPI at H0+24 h and H0+48 h
* Consumption of morphine at H0+24 h and H0+48 h
* Assessment of pain score at 6 months by score ENS at rest , assessment of neuropathic component by DN4 scale. Statement consumption of analgesic treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a lumbar slipped disc surgery
* Aged 18 to 85 years.
* ASA score I-III
* Having given their consent.
* Affiliated with a social security scheme

Exclusion Criteria:

* Patients who must be operated urgently.
* Patients previously operated for lumbar spinal surgery.
* Expected duration of surgery more than 3 hours.
* Severe renal impairment defined by a creatinine clearance less than or equal to 30 mL/min.
* Taking long-term strong opiates .
* Taking long-term corticosteroids or within 48 hours before surgery.
* Taking pregabalin or gabapentin within 48 hours before surgery.
* Drug addiction.
* Patients with cognitive impairment (judged by the investigator) that may interfere with:

informed consent, the collection of endpoints, the use of auto-controlled analgesia.

* Pregnant or nursing women.
* Refusal of the protocol.
* Minor or major protected patients.
* Allergy or other cons-indication to the molecules used in the protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Pain | at H0+2H, at H0+6h, at H0+12h, at H0+24h, at H0+48h
Pain evaluated by ENS during the first mobilization at the edge of the bed | at J0+1 day

SECONDARY OUTCOMES:
Pain | during the first mobilization with standing up at J1
Quality of the standing up (evaluated by Likert scale) | at J0+1day
Patient satisfaction (evaluated by Likert scale) | at J0+1 day
Consumption of morphine | between H0+2h and H0+24h
Pain at rest | at J0+180 days
assessment of neuropathic component DN4 scale | at J0+180 days
statement of analgesic treatment | at J0+180 days
Pain during mobilization | at J0+180 days
Postoperative Nausea and Vomiting | at H0+24h
Postoperative Nausea and Vomiting | at H0+48h
Sedation | at J0 at the arrival in the operating room
Sedation | at J0 at the end of SSPI
Sedation | at H0+24 h
Sedation | at H0+48h
Existence of visual disturbances | at H0, between H0 and H0+48H
Existence of lightheadedness | at H0, between H0 and H0+48H
Existence of urinary retention | at H0, between H0 and H0+48H
Existence of pruritus | at H0, between H0 and H0+48H
Pain | at H0+0h30
pain | at H0+1h
pain | at H0+1h30
pain | at H0+2h
pain | at H0+6h
pain | at H0+12h
pain | at H0+24h
pain | at H0+48h

CONTACTS AND LOCATIONS:
Overall Officials: Bruno VERDIER, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Momon A, Verdier B, Dolomie JO, Gardette M, Pereira B, Curt I, Duale C. A Single Preoperative Administration of Dexamethasone, Low-dose Pregabalin, or a Combination of the 2, in Spinal Surgery, Does Not Provide a Better Analgesia Than a Multimodal Analgesic Protocol Alone. Clin J Pain. 2019 Jul;35(7):594-601. doi: 10.1097/AJP.0000000000000719. PMID 31021886